CLINICAL TRIAL: NCT06012084
Title: The Development and Evaluation of an Internet-delivered Mental Health Prevention Program for Healthy Child Siblings of Individuals With Cystic Fibrosis
Brief Title: The Development and Evaluation of iCF-PWR for Healthy Siblings of Individuals With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Health Authority - Regina Area (Other); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-123
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis; Siblings; Mental Health; Internet-based Intervention
Keywords: cystic fibrosis; siblings; mental health; child; adolescent; sibling relations; Internet-based intervention; anxiety; depression
MeSH Terms: conditions — Cystic Fibrosis; Psychological Well-Being; Anxiety Disorders; Depression | interventions — Health; Health Resources

STUDY DESIGN:
Intervention Model Description: Single-case experimental design (SCED), across-participant AB design. Randomized phase-order will be used in that the start point of the intervention phase will be randomized across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCF-PWR Intervention (Experimental): Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource (iCF-PWR) program is comprised of five text/voice-delivered, animated, interactive modules. The pathways are comprised of the same modules that take approximately 15 to 20 minutes to complete. Modules are comprised of web pages and/or screens with numerous illustrations and interactive components. Written module content will be presented verbally as well as in text format.
  The program modules include: (1) What is CF? (i.e., physiological explanation of CF, prevalence rate); (2) How does my sibling with CF stay healthy? (i.e., review of medication, nutrition, physiotherapy treatment, and why treatment is important); (3) How does CF affect me?; (4) Mental health awareness (i.e., introduction to cognitive behaviour model of emotions-thoughts, feelings, bodily sensations, and behaviours); and (5) Strategies (i.e., ways to challenge unhelpful thoughts, talking about emotions, relaxation).
  Interventions: Behavioral: Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource (iCF-PWR) program

INTERVENTIONS:
Behavioral: Internet-delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource (iCF-PWR) program — The iCF-PWR program is a self-guided mental health prevention program designed for families with CF.

SUMMARY:
The goal of the clinical trial is to test whether a mental health program that is delivered through the Internet works well for healthy children and adolescents with siblings with cystic fibrosis (CF). The main questions it aims to answer are:

* Does the program improve the mental health and quality of life of healthy siblings?
* Does the program improve the relationship between healthy children and adolescents and their sibling with CF?
* Does the program help healthy siblings learn about CF?

Participants will:

* Fill out an online survey asking questions about their family and mental health before the program
* Complete the online mental health program over five weeks
* Fill out a weekly question asking about their mood for 10 weeks
* Fill out an online survey asking questions about their family and mental health after the program

Healthy children and adolescents with siblings with CF will be compared against themselves. Researchers will compare participants scores before starting the program with their scores during and after completing the program. Researchers hope to develop a program that improves mental health, quality of life, sibling relationships, and knowledge about CF.

DETAILED DESCRIPTION:
BACKGROUND: Healthy siblings of individuals with chronic illnesses, such as with cystic fibrosis (CF), have been shown to experience elevated psychological symptoms (e.g., depression, anxiety), negative psychological adjustment, and internalizing behaviours. Psychoeducation, sibling-oriented care, and involvement in siblings' treatments have demonstrated positive outcomes for siblings in terms of psychological wellbeing, social support, and quality of life. At present, there are currently no tailored mental health programs for healthy siblings of individuals with CF. Despite these advances, there is currently no specific mental health program designed for healthy siblings of individuals with CF in Canada. One viable and appealing option for the delivery of mental health services that would eliminate several of the barriers encountered in face-to-face methods of service delivery (e.g., travel to access care, financial restrictions) is through the Internet. Support exists for the effectiveness and efficacy of Internet-delivered psychological treatments for healthy children and children with a range of acute and chronic health conditions. As such, an Internet-delivered method of mental health service delivery designed to target the specific needs of healthy siblings of individuals with CF may be beneficial. The overall goal of the project is to evaluate a recently developed evidence-based, Internet-delivered mental health prevention program for families with CF [called the Internet-Delivered Cystic Fibrosis Mental Health Prevention, Wellness, and Resource program (iCF-PWR)] living in Saskatchewan, that may be helpful in improving mental health and quality of life.

PARTICIPANTS: Six children (aged 8 to 12 years) with CF will be recruited from CF clinics and CF chapters in Canada. Research ethics approval has been approved in those respective health care institutions.

METHODS/PROCEDURES: Preliminary parent consent will be obtained over the phone. A web link (using Qualtrics) to an informed consent/assent form, demographics form, and questionnaires (i.e., measures of CF health, anxiety, depression, health anxiety, anxiety sensitivity, intolerance of uncertainty, quality of life, disease knowledge, and perception of their sibling relationship) will be e-mailed to parent caregiver. The parent caregiver will help facilitate the child's completion of questionnaires online using Qualtrics, a web-based survey software that enables a user-friendly model of conducting surveys. Parents will also complete two questionnaires about the healthy sibling's anxiety, and depression symptoms. Completion of the questionnaires will take approximately one hour. These measures will be completed again upon completion of the program. A link to the post-program questionnaires will be provided via email to parent caregivers to be completed after the program has been completed by the child. Child participants will be also asked to complete a series of one-item ratings of mood and anxiety prior to beginning the program (i.e., phase A) and during completion of the program (i.e., phase B) using Qualtrics. Each phase of the study will be approximately five weeks in length.

Once enrolled, parent caregivers will be provided with a username/password. Participants will be instructed to keep their username/password private. A contact e-mail of the research coordinator will be provided for technical support and instructions on how to operate the site. All contact with participants will be via e-mail, although a telephone number for the research coordinator will also be provided. Supervision of contact with child participants and parent caregivers will be provided by the research supervisor (i.e., Dr. Kristi Wright). Informatics of participant use of the program will be collected (e.g., amount of time spent completing each module, program completion time). Participants will be encouraged to complete one module per week. A reminder e-mail will be sent to parents if their child has not logged onto the program at least once per week. Participants will also be sent email reminders on the days they have been scheduled to complete a rating of mood and anxiety.

ANALYSES: Statistical analyses will be performed using IBM SPSS Statistics-Version 25. Visual analyses are the primary analyses used to determine whether there may be a functional (i.e., three demonstrations of the effectiveness of the intervention effect) or causal relationship between the intervention and the outcome variables. Visual analysis refers to reaching a judgment about the reliability or consistency of an intervention's effects by visually examining the graphed data. The program's effectiveness will be evaluated primarily by examining the changes between baseline (phase A) and post-program (phase B) measures, in addition to changes across the repeated momentary mood and anxiety measure. Baseline and post-program measures and the mood and anxiety ratings will be presented graphically to enable visual inspection. The visual inspection of data will also include analyzing trends in change over time and changes in variability of outcome measures.

If the data suggests a functional or causal relationship may be present, the visual analyses will be supplement with a quantitative analysis method evaluating the magnitude of the intervention effect. Descriptive statistics will be computed for total scores from the outcome measures. Healthy siblings' baseline and post-program total scores from the measure of interest will also be compared to existing community and/or normative data. A series of independent sample t-tests will be computed to compare healthy siblings to similar aged children to assess for potential differences across samples. To evaluate the magnitude of change in outcomes measures from baseline and post-program, a Reliable Change Index (RCI) will be calculated as an indicator of clinically significant change. The RCI will be calculated for each participant by taking their pre-test and post-test total scores and dividing it by the standard error of the difference.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 8 and 12
* have a child or adolescent sibling with cystic fibrosis
* able to speak and read English

Exclusion Criteria:

* have a severe cognitive impairment or a major comorbid medical or psychiatric illness, as this may have interfered with their ability to participate in the program and evaluation process required for the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Mood and Anxiety Rating | 10 Weeks
  Single ratings of self-reported mood and anxiety will be completed ten times over the course of the study. One question will assess mood and one question will assess anxiety using a 3-point Likert scale (0 = none of the time; 1 = some of the time; 2 = a lot of the time) to indicate the frequency of the symptom that day. Ratings will be completed prior to beginning the program (baseline - phase A) and during completion of the program (intervention - phase B). The number of ratings in each phase will vary based on the participant and be distributed equally across the 5-week periods with a minimum of three ratings per phase (i.e., during baseline or intervention).
Change from Baseline in the State-Trait Anxiety Inventory for Children (STAI-C) | Baseline and Week 10 (post-intervention)
  The STAI-C measures general anxiety in children on a continuous scale with items being rated on a 3-point Likert scale reflecting the frequency of anxiety symptom. Total scores can range from a minimum score of 20 to a maximum score of 60.
Change from Baseline in the Children's Depression Inventory-2 (CDI-2) | Baseline and Week 10 (post-intervention)
  The CDI-2 measures cognitive, affective, and behavioural symptoms of depression in children and adolescents on a continuous scale. Each item is rated on a 3-point Likert scale ranging from 0 (absence of symptom) to 2 (definite symptom). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the Childhood Illness Attitudes Scale (CIAS) | Baseline and Week 10 (post-intervention)
  the CIAS assesses fears, beliefs, and attitudes that are associated with health anxiety and abnormal illness behaviour in school children on a continuous scale. Items are rated on a 3-point Likert scale with total scores range from 29 to 87 with higher scores reflecting higher levels of health anxiety associated behaviours.
Change from Baseline in the Childhood Anxiety Sensitivity Index (CASI) | Baseline and Week 10 (post-intervention)
  The CASI measures fear of anxiety-related symptoms in school children on a continuous scale. Each item is rated on a 3-point Likert scale (1 = none; 2 = some; 3 = a lot) with total scores ranging from 18 to 54 and higher scores reflecting higher levels of anxiety sensitivity.
Change from Baseline in the Intolerance of Uncertainty Scale-Revised (IUS-R) | Baseline and Week 10 (post-intervention)
  The IUS-R measures intolerance of uncertainty in children on a continuous scale. Items are rated on a 5-point Likert scale ranging from 1 (not at all like me) to 5 (entirely like me). Total scores range from 12 to 60 with higher scores indicating higher levels of IU.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL-4.0) | Baseline and Week 10 (post-intervention)
  The PedsQL-4.0 measures health-related quality of life in healthy and acute and chronically ill children and adolescents on a continuous scale. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (almost always). The PedsQL-4.0 is comprised of four generic core scales that encompass physical functioning, emotional functioning, social functioning, and school functioning.
Change from Baseline in the Sibling Relationship Questionnaire-Revised (SRQ-R) | Baseline and Week 10 (post-intervention)
  The SRQ-Rdesigned to assess children's perceptions of their siblings in areas of Closeness/Intimacy, Power, Conflict, and Rivalry. On a 5-point Likert scale ranging from 1 (hardly at all) to 5 (extremely much) children are asked to rate how well a characteristic describes their relationship with their sibling. Higher scores on each of the scales and factors indicate greater levels of the specified relationship quality in the sibling relationship.
Change from Baseline in the Disease Knowledge Questionnaire | Baseline and Week 10 (post-intervention)
  The measure was constructed to assess CF disease knowledge as it related to the iCF-PWR content. It is comprised of 13 items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). Higher scores indicate greater CF disease knowledge.

SECONDARY OUTCOMES:
Change from Baseline in the Children's Depression Inventory-2 - Parent Report (CDI-2 P) | Baseline and Week 10 (post-intervention)
  The CDI-2 P assesses a parent's observation of their child's or adolescent's cognitive, affective, and behavioural symptoms of depression. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 2 (much or most of the time). Total raw scores are converted into T-scores with a score of 65 being indicative clinically significant depressive symptoms.
Change from Baseline in the State-Trait Anxiety Inventory - Parent Version (STAI-P) | Baseline and Week 10 (post-intervention)
  The STAI-P assesses state anxiety (i.e., at this present moment) in school children with and without physical symptoms. Items are rated on a 4-point Likert scale reflecting the frequency the anxiety symptom occurs (1 = not at all; 2 = sometimes; 3 = moderately; 4 = very much so). Total scores for the subscales can range from a minimum score of 20 to a maximum score of 80.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi D Wright, Ph.D, Study Director — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow JH, Ellard DR. The psychosocial well-being of children with chronic disease, their parents and siblings: an overview of the research evidence base. Child Care Health Dev. 2006 Jan;32(1):19-31. doi: 10.1111/j.1365-2214.2006.00591.x. PMID 16398788
- [Background] Giallo R, Gavidia-Payne, S. Evaluation of a family-based intervention for siblings of children with disability or chronic illness. Australian e-Journal for the Advancement of Mental Health. 2008; 7(22).
- [Background] Hartling L, Milne A, Tjosvold L, Wrightson D, Gallivan J, Newton AS. A systematic review of interventions to support siblings of children with chronic illness or disability. J Paediatr Child Health. 2014 Oct;50(10):E26-38. doi: 10.1111/j.1440-1754.2010.01771.x. Epub 2010 Jun 27. PMID 20598075
- [Background] Lobato DJ, Kao BT. Integrated sibling-parent group intervention to improve sibling knowledge and adjustment to chronic illness and disability. J Pediatr Psychol. 2002 Dec;27(8):711-6. doi: 10.1093/jpepsy/27.8.711. PMID 12403861
- [Background] O'Haver J, Moore IM, Insel KC, Reed PG, Melnyk BM, Lavoie M. Parental perceptions of risk and protective factors associated with the adaptation of siblings of children with cystic fibrosis. Pediatr Nurs. 2010 Nov-Dec;36(6):284-91; quiz 292. PMID 21291044
- [Background] Quittner AL, Abbott J, Georgiopoulos AM, Goldbeck L, Smith B, Hempstead SE, Marshall B, Sabadosa KA, Elborn S; International Committee on Mental Health; EPOS Trial Study Group. International Committee on Mental Health in Cystic Fibrosis: Cystic Fibrosis Foundation and European Cystic Fibrosis Society consensus statements for screening and treating depression and anxiety. Thorax. 2016 Jan;71(1):26-34. doi: 10.1136/thoraxjnl-2015-207488. Epub 2015 Oct 9. PMID 26452630
- [Background] Gallagher JE, Jackson MA, George MH, Lewtas J. Dose-related differences in DNA adduct levels in rodent tissues following skin application of complex mixtures from air pollution sources. Carcinogenesis. 1990 Jan;11(1):63-8. doi: 10.1093/carcin/11.1.63. PMID 2403860
- [Background] Vermaes IP, van Susante AM, van Bakel HJ. Psychological functioning of siblings in families of children with chronic health conditions: a meta-analysis. J Pediatr Psychol. 2012 Mar;37(2):166-84. doi: 10.1093/jpepsy/jsr081. Epub 2011 Oct 12. PMID 21994420
- [Background] Kazdin AE. Single-case experimental designs. Evaluating interventions in research and clinical practice. Behav Res Ther. 2019 Jun;117:3-17. doi: 10.1016/j.brat.2018.11.015. Epub 2018 Dec 2. PMID 30527785
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127